CLINICAL TRIAL: NCT02222324
Title: A Randomized, Double-Blind, Placebo and Active-Controlled, Single-Dose, 4-Treatment Crossover Study to Evaluate the Effects of E2609 on QTc Interval in Healthy Subjects
Brief Title: A Study to Evaluate the Effects of E2609 on QTc Interval in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: E2609-A001-004
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Subjects
Keywords: QTc Interval; Healthy Subjects
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Treatment B (Experimental): E2609 Low dose
  Interventions: Drug: E2609
- Treatment C (Experimental): E2609 High dose
  Interventions: Drug: E2609
- Treatment D (Active Comparator): Moxifloxacin
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Placebo — 8 placebo tablets matching E2609
  Arms: Treatment A
Drug: E2609 — E2609 will be administered as 8 tablets
  Arms: Treatment B; Treatment C
Drug: Moxifloxacin — Administered as 1 tablet with 7 tablets of placebo matching E2609
  Arms: Treatment D

SUMMARY:
This thorough QT (TQT) study will take place in healthy subjects administered single doses of study drug. It will be a randomized, double-blind, placebo and active-controlled, 4-treatment crossover study. Subjects will be randomized in an equal ratio to one of 12 possible treatment sequences. Each treatment sequence will comprise all 4 treatments.

DETAILED DESCRIPTION:
The study will consist of 2 phases: Prerandomization and Randomization. The Prerandomization Phase will have 2 periods: Screening (up to 27 days) and Baseline Period 1 (1 day). Eligibility will be determined during the Screening Period. The Randomization Phase will consist of 8 periods: Treatment Period 1, Baseline Period 2, Treatment Period 2, Baseline Period 3, Treatment Period 3, Baseline Period 4, Treatment Period 4, and a Follow-Up Period. Each Baseline Period will last 1 day, followed by the corresponding treatment period. On the first day of each treatment period, subjects will receive a single dose of the assigned study drug. During each treatment period, subjects will be required to stay in the clinical unit from the baseline period to 24 hours postdose. Subjects will then be released from the clinic and will undergo a washout interval of at least 13 days, during which time they will return for additional PK sampling.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria to be included in this study:

1. Healthy, non-smoking, male or female subjects ages greater than or equal to 18 years to less than or equal to 55 years old at the time of informed consent
2. Body mass index (BMI) of greater than or equal to 18 to less than or equal to 30 kg/m2 at Screening
3. Females must not be lactating or pregnant at Screening or Baseline (as documented by a negative betahuman chorionic gonadotropin [B-hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
4. Females of childbearing potential must not have had unprotected sexual intercourse within 30 days before study entry and must agree to use a highly effective method of contraception (eg, total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], or have a vasectomized partner with confirmed azoospermia, but not oral contraceptive or contraceptive implant) throughout the entire study period and for 30 days after study drug discontinuation. If currently abstinent, the subject must agree to use a double barrier method as described above if she becomes sexually active during the study period or for 30 days after study drug discontinuation. Hormonal contraceptives (oral or implant) are not permitted forms of contraception in this study. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy or bilateral oophorectomy, all with surgery at least one month before dosing).
5. Male subjects must have had a successful vasectomy (confirmed azoospermia) or they and their female partners must meet the criteria above (ie, not of childbearing potential or practicing highly effective contraception throughout the study period and for 30 days after study drug discontinuation). No sperm donation is allowed during the study period and for 90 days after study drug discontinuation.

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

1. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks before dosing
2. Evidence of disease that may influence the outcome of the study within 4 weeks before dosing (eg, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or subjects who have a congenital abnormality in metabolism)
3. Any history of gastrointestinal surgery that may affect PK profiles of study drugs (eg, hepatectomy, nephrectomy, or digestive organ resection)
4. Any clinically abnormal symptom or organ impairment found by medical history, physical examinations, vital signs, ECG finding, or laboratory test results that requires medical treatment at Screening or Baseline Periods
5. History of any medical condition which, in the opinion of the investigator, may interfere with study procedures or compromise subject safety
6. A prolonged QT/corrected QT interval (QTc) interval (QTc greater than 450 msec) as demonstrated by the mean of triplicate ECGs at Screening or Baseline Periods
7. History of risk factors for torsade de pointes or the use of concomitant medications that prolonged the QT/QTc interval
8. Persistent systolic blood pressure (BP) greater than 130 mmHg or less than 90 mmHg and diastolic BP greater than 85 mmHg or less than 60 mmHg at Screening or Baseline Periods
9. Heart rate less than 50 or greater than 100 beats/minute at Screening or Baseline Periods
10. History of prolonged QT/QTc interval
11. Left bundle branch block at Screening or Baseline Periods
12. History of myocardial infarction or active ischemic heart disease
13. History of clinically significant arrhythmia or uncontrolled arrhythmia
14. Any other clinically significant ECG abnormalities at Screening or Baseline Periods
15. Known history of clinically significant drug allergy (including to study drugs or any of their excipients) at Screening or Baseline
16. Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening or Baseline Periods
17. Active viral hepatitis (B or C) as demonstrated by positive serology at Screening
18. History of drug or alcohol dependency or abuse within the 2 years before Screening, or who have a positive urine drug or alcohol test at Screening or Baseline Periods
19. Use of recreational drugs
20. Intake of caffeinated beverages or food within 72 hours before dosing
21. Intake of nutritional supplements, juice, and herbal preparations or other foods or beverages that may affect the various drug metabolizing enzymes and transporters (eg, alcohol, grapefruit, grapefruit juice, grapefruit-containing beverages, apple or orange juice, vegetables from the mustard green family [eg, kale, broccoli, watercress, collard greens, kohlrabi, brussel sprouts, mustard], and charbroiled meats) within 1 week before dosing
22. Intake of herbal preparations containing St. John's Wort within 4 weeks before dosing
23. Use of prescription drugs within 4 weeks before dosing
24. Intake of over-the-counter (OTC) medications within 2 weeks before dosing
25. Smoking or use of tobacco or nicotine-containing products within 4 weeks before dosing
26. Engagement in strenuous exercise within 2 weeks before dosing (eg, marathon runners, weight lifters)
27. Currently enrolled in another clinical trial or used any investigational drug or device within 30 days preceding informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QTcF obtained from ECGs extracted from the Holter recordings | Up to 24 hours postdose during each treatment period
  Holter recordings are taken from a portable device for continuously monitoring various electrical activity of the cardiovascular system for at least 24 hours. Baseline is defined as the mean of predose QTcF values obtained from ECGs extracted from Holter recordings before dosing during each treatment period.

SECONDARY OUTCOMES:
Change from baseline in ECG recordings: PR interval | Predose and then up to 24 hours postdose in each treatment period
  Electrocardiograms will be extracted from the continuous digital recording at 3 predose time points. Other time points may be evaluated as well.
Change from baseline in ECG recordings: QRS interval | Predose and then up to 24 hours postdose in each treatment period
  Electrocardiograms will be extracted from the continuous digital recording at 3 predose time points. Other time points may be evaluated as well.
Change from baseline in ECG recordings: HR | Predose and then up 24 hours postdose in each treatment period
  Electrocardiograms will be extracted from the continuous digital recording at 3 predose time points. Other time points may be evaluated as well.
Change from baseline in ECG recordings: RR interval | Predose and then at up to 24 hours postdose in each treatment period
  Electrocardiograms will be extracted from the continuous digital recording at 3 predose time points. Other time points may be evaluated as well.
Change from baseline in ECG recordings: T wave morphology | Predose and then at up to 24 hours postdose in each treatment period
  Electrocardiograms will be extracted from the continuous digital recording at 3 predose time points. Other time points may be evaluated as well.
Pharmacokinetics of E2609: Cmax | Up to 84 Days
  Maximum drug concentration
Pharmacokinetics of E2609: tmax | Up to 84 Days
  Ttime to reach maximum (peak) concentration following drug administration
Pharmacokinetics of E2609: AUC(0-t) | Up to 84 Days
  Area under the concentration x time curve from time = 0 to time of last measurable concentration
Pharmacokinetics of E2609: AUC(0-72h) | Up to 84 Days
  Area under the concentration x time curve from time = 0 to 72 hours postdose
Pharmacokinetics of E2609: AUC(0-inf) | Up to 84 Days
  Area under the concentration x time curve from time = 0 to infinity
Pharmacokinetics of E2609: t1/2 | Up to 84 Days
  Terminal elimination half-life
Pharmacokinetics of E2609: CL/F | Up to 84 Days
  Apparent total clearance following extravascular administration
Pharmacokinetics of E2609: Vz/F | Up to 84 Days
  Apparent volume of distribution following extravascular administration

CONTACTS AND LOCATIONS:
Locations (1):
- San Antonio, Texas, United States